CLINICAL TRIAL: NCT05673239
Title: Effects of L-carnitine Therapy on the Heart of Maintenance Hemodialysis Patients: A Multicenter, Prospective, Non-randomized, Controlled Real-world Study
Brief Title: Effects of L-carnitine Therapy on the Heart of Maintenance Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-ZKNT-001
Record Dates: First submitted 2022-11-29; First posted 2023-01-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2023-01

CONDITIONS: Renal Dialysis
Keywords: Renal Dialysis; Cardiac Function Tests; real-world study; multicenter; prospective; non-randomized; controlled
MeSH Terms: interventions — Carnitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Experimental): The patients in the test group were injected with levocarnitine on each dialysis day, and other conventional treatment drugs such as hemodialysis drugs were maintained in the original scheme and recorded in detail on the CRF form.
  Interventions: Drug: Levocarnitine Injection
- Control group (No Intervention): The patients in the control group were the same as those in the test group, except that they were not treated with L-carnitine.

INTERVENTIONS:
Drug: Levocarnitine Injection — The patients in the test group were injected with 1-2g (10-20mg/kg) levocarnitine on each dialysis day
  Arms: Test group

SUMMARY:
This study is intended to be a multicenter, prospective, non-randomized, controlled real-world study. Patients receiving L-carnitine injection were included in the experimental group and the control group according to whether they received L-carnitine injection. Patients receiving L-carnitine injection were included in the experimental group, and those receiving L-carnitine injection were included in the control group.To observe the effects of L-carnitine on cardiac function in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Maintenance hemodialysis patients;
* 18 years<80 years;
* Have clear consciousness and independent behavior ability;
* Before dialysis, the total carnitine concentration was less than 40 umol/L, or the free carnitine concentration was less than 35 umol/L.

Exclusion Criteria:

* Acute cardiovascular and cerebrovascular diseases occurred within 1 month;
* Infectious diseases occurred within 1 month; Treatment with glucocorticoid or immunosuppressant;
* Patients who have used L-carnitine within 2 weeks.
* Hematological system tumor or tumor;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1008 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Left ventricular ejection fraction | baseline and week 12

SECONDARY OUTCOMES:
Change from baseline in Brain natriuretic peptide level | baseline ,week 4 and week 12
Change from baseline in left ventricular short axis shortening rate | baseline and week 12
Change from baseline in stroke volume | baseline and week 12
Change from baseline in the ratio of peak E to peak A of mitral valve blood flow velocity in early and late diastolic periods | baseline and week 12
Change from baseline in serum albumin | baseline and week 12
Change from baseline in upper arm circumference | baseline and week 12
Change from baseline in prealbumin | baseline and week 12
Change from baseline in hemoglobin | baseline and week 12

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No